CLINICAL TRIAL: NCT02958579
Title: A Population Based Cohort Study on Metabolic Syndrome Complications, and Mortality; (MetSCoM) Study
Brief Title: a Population Based Study on Metabolic Syndrome Complications, and Mortality
Acronym: MetSCoM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 95-03-191-33053; 957275 (Other Grant/Funding Number: National Institute for Medical Research Development (NIMAD))
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Obesity: Body mass index (BMI) score > 25.2 kg/m2 for women and > 27.3 kg/m2 for men or Waist circumference > 90 cm
  Interventions: Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.
- Pre-diabetics or diabetics: if any of followings is identified the participant is regarded as diabetics and will be recruited in this arm;
  1. Fasting Plasma glucose (FPG) level ≥ 7.0 mmol/l (126 mg/dL)
  2. Plasma glucose ≥ 11.1 mmol/l (200 mg/dL) two hours after a 75 g oral glucose load as in a glucose tolerance test
  3. Symptoms of hyperglycemia and casual plasma glucose ≥ 11.1 mmol/l (200 mg/dL)
  4. Glycated hemoglobin (A1C) ≥ 6.5% if any of followings is identified the participant is regarded as pre-diabetics and will be recruited in this arm;
  1- FPG levels of 100-125 mg/dl (5.6-6.9 mmol/l). 2-Two-h plasma glucose (2HPP) in the 75 g oral glucose tolerance test of 140-199 mg/dl (7.8- 11.0 mmol/l)
  Interventions: Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.
- Hypertension: Systolic blood pressure (SBP) ≥ 130mmHgand/or diastolic blood pressure (DBP) ≥ 85mmHg or use of anti-hypertensive drugs
  Interventions: Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.
- hypertriglyceridemia: Serum triglyceride ≥150 mg/dL
  Interventions: Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.
- Low high density lipoprotein -cholesterol (HDL-c): Serum HDL-C of <40 mg/dL for men, <50 mg/dL for women,
  Interventions: Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.

INTERVENTIONS:
Other: No intervention will be done. Participants are on standard care and the treatments will be recorded because of observational nature of this study.

SUMMARY:
Metabolic syndrome (MetS) is recognized as clustering of a number of components including hypertension, hypertriglyceridemia, low serum high-density lipoprotein cholesterol (HDL-C), impaired glucose metabolism (IGM), and abdominal obesity. It has been tightly linked to thrombotic vascular events including coronary heart disease (CHD). Worldwide prevalence of MetS is on the rise. People living in Iran, a country located in the Middle-East region, have distinct behavioral, environmental and social exposures which certainly affect the prevalence and incidence of metabolic syndrome and its comorbidities.We hypothesized that these factors may affect the course of metabolic syndrome and the burden that it imposes to the community. The purposes of MetSCoM are as follows;

1. To find the incidence of T2D, microvascular complications of T2D (diabetic retinopathy, diabetic neuropathy and diabetic kidney disease), CVD, and mortality rate of subjects metabolic syndrome.
2. To find the association of baseline, mean value during follow up visits and visit to visit variability in anthropometric variables and several metabolic laboratory variables with metabolic syndrome and its complications.
3. To find the effect of behavioral variables and environmental exposures on the course of metabolic syndrome.
4. To identify the best anthropometric, laboratory, life-style and environmental predictors of CVD and mortality rate in subjects with metabolic syndrome.
5. To estimate the economic burden of metabolic syndrome and its related

DETAILED DESCRIPTION:
A biphasic observational study will be conducted on participants with any component of metabolic syndrome in Tehran, Iran. Phase one of the study is a cross-sectional study, while the second phase is a prospective cohort. In phase one of study, the prevalence of any metabolic disorder will be estimated in the study population and the association of biochemical variables, behavioral and environmental variables with each metabolic disorder will be investigated. Afterwards, through the phase two, those with any component of metabolic syndrome will be followed to record the incidence of diabetes, vascular complications of diabetes, non-alcoholic fatty liver disease, (NAFLD), cancers, mortality rate and finally estimation of economic burden of metabolic syndrome and its components in study population. Participants will be recruited from four health surveillance centers located at East, West, North and South of Tehran, the capital city of Iran. The latitude of Tehran is 35°41' North, and 51°25' East. Participants will be followed for at least 10 years and we plan to extend this time if possible. Anthropometric, biochemical, behavioral and meteorological measurements will done on scheduled timeline.

ELIGIBILITY:
Inclusion Criteria:

* Obesity or central obesity, or
* Diabetes (Fasting Plasma glucose (FPG) level ≥ 7.0 mmol/l (126 mg/dL), or Plasma glucose ≥ 11.1 mmol/l (200 mg/dL) two hours after a 75 g oral glucose load as in a glucose tolerance test, or Symptoms of hyperglycemia and casual plasma glucose ≥ 11.1 mmol/l (200 mg/dL), or Glycated hemoglobin (A1C) ≥ 6.5%),
* pre-diabetes (FPG levels of 100-125 mg/dl (5.6-6.9 mmol/l), or 2-h plasma glucose (2HPP) in the 75 g oral glucose tolerance test of 140-199 mg/dl (7.8-11.0 mmol/l), or
* Hypertension (Systolic blood pressure (SBP) ≥ 130mmHgand/or diastolic blood pressure (DBP) ≥ 85mmHg or use of anti-hypertensive drugs), or
* Low HDL-c (Serum HDL-C of <40 mg/dL for men, <50 mg/dL for women,)
* Hypertriglyceridemia, (TG>150 mg/dL)

Exclusion Criteria:

* type 1 diabetes
* type 2 diabetes who required insulin therapy at baseline
* gestational diabetes
* Any malignancy, rheumatologic diseases, chronic kidney, lung or heart diseases at baseline at baseline
* known hepatitis due to infectious and auto-immune diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All community dwellers aged greater than 40 years who are willing to participate will be included if met any of the following eligibility criteria; (1) central obesity, or (2) obesity, or (3) T2D or prediabetes, or (4) hypertension, or (5) hypertriglyceridemia, or (6) low high density lipoprotein-cholesterol (HDL-C).
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2005-01; Primary Completion 2017-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
incidence of CVD | 10 years
incidence of microvascular complications of T2D (diabetic retinopathy, diabetic neuropathy, diabetic kidney disease), and diabetic foot | 10 years
incidence of non-alcoholic fatty liver disease (NAFLD) | 10 years
incidence of colorectal, breast and cervical cancers | 10 years
mortality rate | 10 years

SECONDARY OUTCOMES:
economic burden of metabolic syndrome | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Afarideh, MD, MPH, Principal Investigator — Tehran University of Medical Sciences; Alireza Ghajar, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Result] Heidari B, Nargesi AA, Hafezi-Nejad N, Sheikhbahaei S, Pajouhi A, Nakhjavani M, Esteghamati A. Assessment of serum 25-hydroxy vitamin D improves coronary heart disease risk stratification in patients with type 2 diabetes. Am Heart J. 2015 Sep;170(3):573-9.e5. doi: 10.1016/j.ahj.2015.06.017. Epub 2015 Jun 27. PMID 26385042
- [Result] Afarideh M, Aryan Z, Ghajar A, Noshad S, Nakhjavani M, Baber U, Mechanick JI, Esteghamati A. Complex association of serum alanine aminotransferase with the risk of future cardiovascular disease in type 2 diabetes. Atherosclerosis. 2016 Nov;254:42-51. doi: 10.1016/j.atherosclerosis.2016.09.009. Epub 2016 Sep 9. PMID 27684605
- [Result] Nargesi AA, Heidari B, Esteghamati S, Hafezi-Nejad N, Sheikhbahaei S, Pajouhi A, Nakhjavani M, Esteghamati A. Contribution of vitamin D deficiency to the risk of coronary heart disease in subjects with essential hypertension. Atherosclerosis. 2016 Jan;244:165-71. doi: 10.1016/j.atherosclerosis.2015.11.020. Epub 2015 Nov 23. PMID 26647372
- [Result] Aryan Z, Noshad S, Afarideh M, Esteghamati A. Comment on Sharif et al. HDL Cholesterol as a Residual Risk Factor for Vascular Events and All-Cause Mortality in Patients With Type 2 Diabetes. Diabetes Care 2016;39:1424-1430. Diabetes Care. 2016 Oct;39(10):e189. doi: 10.2337/dc16-1211. No abstract available. PMID 27660132
- [Result] Afarideh M, Noshad S, Ghajar A, Aryan Z, Khajeh E, Hosseini Shirvani S, Bonnet F, Esteghamati A. Family history of diabetes and the risk of coronary heart disease in people with or without type 2 diabetes. Diabetes Metab. 2017 Apr;43(2):180-183. doi: 10.1016/j.diabet.2016.07.032. Epub 2016 Sep 17. No abstract available. PMID 27644597
- [Result] Faghihi-Kashani S, Bonnet F, Hafezi-Nejad N, Heidari B, Aghajani Nargesi A, Sheikhbahaei S, Ebadi M, Esteghamati A. Fasting hyperinsulinaemia and 2-h glycaemia predict coronary heart disease in patients with type 2 diabetes. Diabetes Metab. 2016 Feb;42(1):55-61. doi: 10.1016/j.diabet.2015.10.001. Epub 2015 Oct 31. PMID 26531321
- [Result] Esteghamati A, Hafezi-Nejad N, Zandieh A, Sheikhbahaei S, Ebadi M, Nakhjavani M. Homocysteine and metabolic syndrome: from clustering to additional utility in prediction of coronary heart disease. J Cardiol. 2014 Oct;64(4):290-6. doi: 10.1016/j.jjcc.2014.02.001. Epub 2014 Mar 14. PMID 24631466
- [Result] Esteghamati A, Hafezi-Nejad N, Sheikhbahaei S, Heidari B, Zandieh A, Ebadi M, Nakhjavani M. Risk of coronary heart disease associated with metabolic syndrome and its individual components in Iranian subjects: a matched cohort study. J Clin Lipidol. 2014 May-Jun;8(3):279-86. doi: 10.1016/j.jacl.2014.02.002. Epub 2014 Feb 15. PMID 24793349
- [Result] Sheikhbahaei S, Fotouhi A, Hafezi-Nejad N, Nakhjavani M, Esteghamati A. Serum uric acid, the metabolic syndrome, and the risk of chronic kidney disease in patients with type 2 diabetes. Metab Syndr Relat Disord. 2014 Mar;12(2):102-9. doi: 10.1089/met.2013.0119. Epub 2014 Jan 21. PMID 24447037
- [Derived] Aryan Z, Ghajar A, Faghihi-Kashani S, Afarideh M, Nakhjavani M, Esteghamati A. Baseline High-Sensitivity C-Reactive Protein Predicts Macrovascular and Microvascular Complications of Type 2 Diabetes: A Population-Based Study. Ann Nutr Metab. 2018;72(4):287-295. doi: 10.1159/000488537. Epub 2018 Apr 25. PMID 29694948